CLINICAL TRIAL: NCT01317472
Title: A Double-Blinded, Placebo-Controlled Trial to Investigate Dexlansoprazole for the Treatment of Laryngopharyngeal Reflux
Brief Title: The Effects of Dexlansoprazole for the Treatment of Throat-Related Reflux
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left institution
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSA-NC-DEX-115
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Laryngopharyngeal Reflux
Keywords: laryngopharyngeal reflux, acid reflux, throat reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexlansoprazole (Experimental): Patients who agree to participate in the study will be randomized to receive 60 mg po QAM Kapidex (1 hour AC).
  Interventions: Drug: dexlansoprazole
- Sugar pill (Placebo Comparator): Patients who agree to participate in the study will be randomized to receive 60 mg po QAM Kapidex (1 hour AC) or 1 tablet of placebo QAM (1 hour AC).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dexlansoprazole — 60 mg dexlansoprazole QAM (1 hour AC) for 2 months
  Other Names: Dexilant
  Arms: Dexlansoprazole
Drug: Placebo — 1 tablet of placebo QAM (1 hour AC) for 2 months
  Arms: Sugar pill

SUMMARY:
Recent studies have demonstrated that patients with throat-related reflux often require twice daily proton pump inhibitor therapy to attain significant symptomatic improvement, with once daily therapy offering little relief. As dexlansoprazole is a twice-daily release proton pump inhibitor requiring only once-daily dosing, it may provide laryngopharyngeal reflux (LPR) symptomatic relief comparable to that of twice daily dosing, yet be more readily approved by third party payers because of its once daily dosing requirements. It is hypothesized that, in patients with pharyngeal-probe proven throat reflux, there will be significantly greater improvement in symptoms and pharyngeal probe findings in those patients receiving dexlansoprazole than those receiving placebo alone.

DETAILED DESCRIPTION:
The aim of the study is to compare outcomes, based on RSI-based symptomatic improvement and pharyngeal probe results, after LPR patients are treated for two months with once-daily (QAM) Kapidex versus placebo.Forty patients with pharyngeal pH probe-documented LPR and an elevated reflux symptom index (RSI) (≥14) will be enrolled into a double-blinded placebo controlled study. Twenty patients will receive Kapidex once daily, while twenty receive placebo. Patients will return at two months for evaluation with repeat RSI documentation and repeat pharyngeal pH probe testing. Student t-test will be used to determine if the change in RSI and pH-probe results differs between the study and placebo group.

ELIGIBILITY:
Inclusion Criteria:patients with an abnormal Restech pH probe study and also have an RSI of 14 or greater will be invited to participate in the study

Exclusion Criteria:known intolerance or allergy to proton pump inhibitors, hypersecretory conditions (Zollinger-Ellison), self-reported anxiety/depression (shown to affect RSI),16 history of laryngeal irradiation, or have been on twice daily Proton pump inhibitors (PPI) therapy for greater than 2 months without symptomatic relief (with an RSI ≥14)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Halum, MD, Principal Investigator — Indiana University
Locations (1):
- Clarian North Hospital -- IUMG Clinic, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Pill: Patients who agree to participate in the study will be randomized to receive 60 mg po QAM Kapidex (1 hour AC) or 1 tablet of placebo QAM (1 hour AC).
  dexlansoprazole: 60 mg dexlansoprazole QAM (1 hour AC) for 2 months
Period: Overall Study
Arm/Group | Dexlansoprazole | Sugar Pill
Started | 9 | 2
Completed | 7 | 2
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unrelated hospitalization | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole | Sugar Pill | Total
Number analyzed (Participants) | 9 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Reflux Symptom Index (RSI)
Description: The Reflux Symptom Index (RSI) is a 9-item measure with each symptom rated from 0 (no problem) to 5 (severe problem), for a total possible range of 0 (no problem) to 45 (severe problem). An RSI of >13 is considered to be abnormal.
Time Frame: Baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole | Sugar Pill
Number analyzed (Participants) | 7 | 2
units on a scale | 18 (3.95) | 13 (4.54)

ADVERSE EVENTS:
Arm/Group | Dexlansoprazole | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 0/9 | 0/2

LIMITATIONS AND CAVEATS:
very poor recruitment. patients were not willing to enter study because they did not want to take a chance on receiving placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No